CLINICAL TRIAL: NCT05834829
Title: Investigation of Low-intensity Focused Ultrasound to the Salience Network on Autonomic Function
Brief Title: Low-intensity Focused Ultrasound and Autonomic Response
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 23-049
Record Dates: First submitted 2023-01-12; First posted 2023-04-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Autonomic Dysfunction
MeSH Terms: conditions — Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: three arm model, participants receive each intervention/sham (dPI, ACC, or Sham) one per study visit in a randomized order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham application during a single randomized session (1 of 3 sessions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- dPI (Experimental): LIFU to the dPI
  Interventions: Device: Low-intensity focused ultrasound neuromodulation
- ACC (Experimental): LIFU to the ACC
  Interventions: Device: Low-intensity focused ultrasound neuromodulation
- Sham (Sham Comparator): Sham LIFU application
  Interventions: Device: Sham Low-intensity focused ultrasound

INTERVENTIONS:
Device: Low-intensity focused ultrasound neuromodulation — ultrasound transducer applying low intensity waveforms to targeted brain regions for neuromodulation.
  Arms: ACC; dPI
Device: Sham Low-intensity focused ultrasound — sham application of ultrasound using blocking of the ultrasound waves of the transducer.
  Arms: Sham

SUMMARY:
Studying the effects of Low Intensity Focused Ultrasound (LIFU) to the dorsal posterior insula (dPI) and dorsal anterior cingulate cortex (dACC) on autonomic control using a test to probe the autonomic system. A cold pressor task will be performed pre and post LIFU application. Physiologic recordings will be recorded throughout.

DETAILED DESCRIPTION:
Characterize the effect of LIFU to the bilateral dorsal posterior insula (dPI) and dorsal anterior cingulate cortex (dACC)) on autonomic control. The dPI is a critical brain area involved in autonomic function, being a core recipient of ascending pain and autonomic function. Similarly, the dACC has been strongly implicated in autonomic control and works with the insula for autonomic processing. Inconveniently, these brain regions lie deep to the cortex, prohibiting access using conventional noninvasive methods like transcranial magnetic stimulation (TMS). LIFU can be focused at depth to reach the insula and ACC with high spatial precision. However, the effect of LIFU to the human dPI and dACC on autonomic control is unknown. To address this, the investigators will target the right dPI and the dACC to assess how LIFU to each of these areas affects autonomic responses and subjective report to the cold pressor task, a safe, reproducible autonomic challenge.

ELIGIBILITY:
Inclusion Criteria:

* Does not meet exclusion criteria.

Exclusion Criteria:

The exclusion criteria below are regularly implemented in MRI, CT, and EEG experiments for the safety of the subjects and for data quality assurance.

* Claustrophobia (scanning environment may be uncomfortable).
* Contraindications to MRI: including pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
* Contraindications to CT: pregnancy
* Active medical disorder or treatment with potential central nervous system (CNS) effects (e.g. Alzheimer's) -
* History of neurologic disorder. (e.g. Parkinson's, Epilepsy, or Essential Tremor)
* History of head injury resulting in loss of consciousness for >10 minutes.
* History of alcohol or drug dependence (through self-report).
* History of cardiac disease
* A current or prior use of any cardiac medication (e.g. beta blockers or other anti-arrhythmics)
* A history of diabetes mellitus or use of diabetic medications (e.g. metformin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sympathetic tone response - Heart Rate Variability (HRV) | through study completion, an average of 1 month
  Changes in HRV
Sympathetic tone response - Heart Rate (HR) | through study completion, an average of 1 month
  Changes in HR
Sympathetic tone response - Blood Pressure (BP) | through study completion, an average of 1 month
  Changes in BP (systolic and diastolic pressure)
Sympathetic tone response - Electrodermal Response (EDR) | through study completion, an average of 1 month
  Changes in EDR
Sympathetic tone response - Electroencephalography (EEG) | through study completion, an average of 1 month
  Changes in low and high frequency power

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No